CLINICAL TRIAL: NCT04292080
Title: Long-Term Analysis of DImethyl Fumarate, to Slow the Growth of Areas of Geographic Atrophy
Acronym: LADIGAGA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P170919; 2019-003413-33 (EudraCT Number); 2024-510741-33-00 (EU CTIS Number)
Record Dates: First submitted 2020-02-17; First posted 2020-03-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Dimethyl Fumarate

STUDY DESIGN:
Intervention Model Description: Participants receive an intervention throughout the protocol. There are 2 groups :
  Group 1 : Group TECFIDERA
  Group 2 : No active (No treatment)
Masking Description: No masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TECFIDERA™ (Experimental): Patients will receive oral administration of Dimethyl Fumarate (Tecfidera™) 120 mg twice a day for the first week and then 240 mg of Tecfidera twice a day for 51 weeks following approved standard treatment scheme.
  Interventions: Drug: Dimethyl Fumarate (TECFIDERA™)
- No comparator (Other): Patients will receive no specific treatment (standard of care) up to 24 months following randomization.
  Interventions: Other: No active : no treatment

INTERVENTIONS:
Drug: Dimethyl Fumarate (TECFIDERA™) — Dimethyl fumarate is a white to off-white powder that is highly soluble in water with a molecular mass of 144.13, containing 120 mg or 240 mg of dimethyl fumarate The starting dose for TECFIDERA is 120 mg twice a day orally. After 7 days, the dose should be increased to the maintenance dose of 240 mg twice a day orally. Body weight, gender, and age do not require dosage adjustment.
  Arms: Group TECFIDERA™
Other: No active : no treatment — Patients will receive no specific treatment (standard of care) up to 24 months following randomization.
  Arms: No comparator

SUMMARY:
The primary objectives of the study are to assess the safety, tolerability and evidence of activity of 12 months oral treatment with TEFIDERA® in subjects with Geographic Atrophy associated with Age-Related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
Age-related Macular Degeneration (AMD) is the leading cause of irreversible blindness in the industrialized world. Approximately 80% of patients with AMD suffer from the dry form of the disease also called geographic atrophy (GA) which is characterized by the progressive loss of photoreceptors and RPE that are essential to the visual cycle. There is currently no therapy to cure GA. This represent a major health problem with millions patients worldwide.

GA is a complex multifactorial disease influenced by: aging, environmental factors, genetic predispositions, oxidative stress and inflammation. Oxidative stress is the major environmental risk factor of developing AMD. Whereas inflammation, is now, recognized as one of the main player in AMD pathophysiology. Therefore, antioxidant and immunosuppressive therapies are susceptible to be beneficial in humans for patients with GA.

Dimethyl Fumarate activates the NRF2 pathway, which is the major transcription factor regulating anti-oxidative enzymes production. Dimethyl Fumarate commercialized under the name TECFIDERA® by BIOGEN is an effective antioxidant and immunosuppressive drug, used to treat patients with Multiple Sclerosis (MS), an autoimmune disease of the Central Nervous System leading to progressive disability. This new therapeutic agent may be easily repurposed to treat GA patients and could reduce or slow photoreceptors and RPE degeneration and the associated vision loss.

In this randomized, open labelled trial we will evaluate the safety and efficacy of TECFIDERA®, in two groups of patients (treated vs. untreated) with GA. This is the first time this strategy, based on evidences that oxidative stress and inflammation are central in GA physiopathology, will be tested in patients with dry AMD.

ELIGIBILITY:
Inclusion Criteria:

Age 55 years of age to 85 years old at the moment of inclusion

* Participant must understand and sign the protocol's informed consent document
* Participant must have central or non-central geographic atrophy (GA) in at least one eye. GA should be at least 0.75 disk areas (DA) in size but no more than 8 disk areas (DA); approximately 2.54 mm2 is 1 DA. (GA is defined as one or more well-defined, usually more or less circular patches of partial or complete de-pigmentation of the retinal pigment epithelium (RPE), typically with exposure of underlying choroïdal blood vessels. Even if much of the RPE appears to be preserved and large choroïdal vessels are not visible, a round patch of RPE partial de-pigmentation may still be classified as early GA. If a patient has 2 eligible eyes; one eye will be the "study eye", graded and evaluated during the whole duration of the study)
* Participant must have a steady fixation in the study eye in the foveal or parafoveal area and media clear enough for good quality photographs
* Participant must have visual acuity between 20/20 and 20/200 in the affected eye
* No suggestive sign of progressive multifocal leukoencephalopathy on brain MR Imaging within 3 months of Tecfidera© treatment Initiation (Only the patients randomized in the TECFIDERA Group will have to go through the MR Imaging)
* Male participants with female partners capable of conceiving children will be required to use contraception (condom) during the study and for four months after their last experimental treatment caps
* No documented history of heart disease, absence of family history of sudden death, and QTc duration within normal value (<480ms)
* Participants must be affiliated to a social security scheme

Exclusion Criteria:

* Participant is in another interventional investigational study < 3 months before inclusion
* Participant is unable to comply with study procedures or follow-up visits
* Participant has evidence of ocular disease other than GA in either eye that may confound the outcome of the study (e.g., glaucoma, diabetic retinopathy with 10 or more hemorrhages or micro-aneurysms, uveitis, pseudo-vitelliform macular degeneration, exudative macular degeneration, moderate/severe myopia)
* Participant with antecedent of neo-vascular AMD.
* Participant has received treatment for exudative AMD, such as macular laser, photodynamic therapy (PDT) or anti-vascular endothelial growth factor (anti-VEGF) therapy intra-vitreal (IVT) injection or of any agent (e.g., triamcinolone) in the study eye within the last four months prior to study enrollment. Vitamin supplementation for AMD is not considered an exclusionary criterion
* Participant has had a vitrectomy in the study eye
* Participant is expected to need ocular surgery during the course of the trial
* Participant has undergone lens removal in the last three months or Yttrium Aluminium Garnet (YAG) laser capsulotomy within the last month
* Participant is on chemotherapy
* Participant is on chronic (more than 3 months) immunosuppressive medication administered via ocular or systemic route(s) or is immunosuppressed
* Participant is on ocular or systemic medications known to be toxic to the lens, retina or optic nerve
* Participant with a history of malignancy that would compromise the 2-year study survival
* Participant with a history of ocular herpes simplex virus (HSV)
* Contra-indications or known hyper-sensibility to Dimethyl Fumarate (Tecfidera™) or experimental treatment excipients
* Severe active gastrointestinal disease
* Contra-indications to an MRI using gadolinium such as pace maker, cardiac valve non IRM compatible, cochlear implant or any metallic implant non IRM compatible.
* Any contraindications to gadolinium including pregnancy, previous allergic reaction, severe kidney disease
* Any contraindications to aspirin
* Any screening laboratory value (hematology, serum chemistry or urinalysis) 3 times above normal values or that in the opinion of the Investigator is clinically significant and not suitable for study participation
* Lymphopenia below normal laboratory values at inclusion.
* Severe impairment of a vital organ including severe liver and renal impairment
* Previous organ allograft
* Patients taking the following non-authorized treatment 3 months prior enrolment: other fumaric acid derivatives (topical occular or systemic), immuno-modulators via ocular or systemic routes (including interferons, sirolimus, chronic use of glucocorticoids) cytotoxic treatments and live attenuated vaccines.(NB: During the experimental treatment period and 3 months thereafter the concomitant use of non-authorized treatment cited above is not allowed in patients randomized in the TEFIDERA group)
* Patients taking the following non-authorized treatment 3 months prior enrolment: nephrotoxic treatment (aminoglycosides, diuretics, nonsteroidal anti-inflammatory drugs (via ocular or systemic routes) or lithium). (NB: During the experimental treatment period and 3 months thereafter the concomitant use of non-authorized nephrotoxic treatment cited above is not allowed in patients randomized in the TEFIDERA group)
* Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control)
* History of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years that could be worsened by immunosuppression (In case of history of cancer the risk of immunosuppression must be determined by a specific oncology consultation prior to enrollment.)
* Ocular or peri-ocular inflammation or infection in either eye
* Presence of active or inactive toxoplasmosis in any or both eye(s)
* Presence of active or latent tuberculosis infection
* Female participants of child bearing potential (those who are not post-menopausal or surgically sterile). Postmenopausal state is 12 months of amenorrhea + high level of FSH if required.
* Persons under curatorship or guardianship

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2029-04-07 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Month 12 in total area of GA Lesion(s) in the study eye (in mm2) as Measured by Fundus Autofluorescence (FAF) | 12 Months

SECONDARY OUTCOMES:
Incidence and severity of ocular and systemic treatment-related adverse events as assessed by CTCAE v4.0". | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric SOUIED, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre intercommunal de Créteil, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No